CLINICAL TRIAL: NCT05153811
Title: Novel Extensions of Alcohol Contingency Management in People Living With HIV
Brief Title: The Less is More Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: University of Miami (Other); University of Louisville (Other); Florida State University (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CED000000577; P01AA029543 (NIH); PRO00035889 (Other: UFirst); OCR41499 (Other: UF OnCore); CED000000577 (Other: UF IRB Number)
Record Dates: First submitted 2021-12-02; First posted 2021-12-10 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Use
MeSH Terms: conditions — Alcohol Drinking | interventions — Counseling; Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-Contingent Condition (Experimental): Participants will wear a wrist biosensor with daily CM based on smartphone breathalyzer readings for 30 days; then for a second 30 days, encouragement to reduce drinking but payment not based on drinking.
  Interventions: Behavioral: Counseling
- mHealth and CM (Experimental): Participants will wear a wrist biosensor with daily CM based on smartphone breathalyzer readings for 30 days; then for a second 30 days, weekly CM based on wrist biosensor readings. Participants will also interact with a mobile health application to facilitate drinking reduction.
  Interventions: Behavioral: Counseling; Behavioral: mHealth
- CM (Experimental): Participants will wear a wrist biosensor with daily CM based on smartphone breathalyzer readings for 30 days; then for a second 30 days, weekly CM based on wrist biosensor readings
  Interventions: Behavioral: Counseling

INTERVENTIONS:
Behavioral: Counseling — Brief counseling including personalized feedback on breath alcohol concentration, cognitive task performance and physical functioning
  Arms: CM; mHealth and CM
Behavioral: mHealth — Participants will engage with an application designed to gamify drinking reduction.
  Arms: mHealth and CM
Behavioral: Counseling — Brief counseling including personalized feedback on breath alcohol concentration, cognitive task performance and physical functioning.
  Arms: Non-Contingent Condition

SUMMARY:
In this project, the investigators will implement innovations to extend use of Contingency Management (CM) to facilitate alcohol use reduction among people living with HIV (PLWH). The investigators' approach to extending CM will use mobile health (mHealth) tools including a smartphone breathalyzer device with accompanying app and a wrist worn alcohol biosensor. Participants will be engaged in mobile facilitated CM for 30-60 days with follow-up out to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Frequent alcohol use in the past 30 days based on responses on the Timeline Followback (TLFB; Sobell and Sobell, 2003)
* HIV positive
* Fluency in English
* Willingness to attempt alcohol abstinence for at least 30 days and then to attempt alcohol use on fewer days than at baseline after that
* Willingness to use smartphone applications and biosensor devices (i.e., breathalyzer device and wrist sensor) for alcohol use reduction purposes in the study. If participants do not have a compatible smartphone to use, they will be loaned one by the study

Exclusion Criteria:

* Psychiatric conditions that would interfere with participation in the study
* Current alcohol withdrawal as indicated by a score of 8 or higher on the Clinical Institute Withdrawal Scale (CIWA; Sullivan et al., 1989) or lifetime history of medically assisted detoxification
* Two positive breath alcohol concentration (BrAC) readings (i.e., > 0.00%) at an in-person screening appointment. After participants blow their first positive BrAC, they will be allowed to reschedule and participate at another time, however if they blow a second positive BrAC, they will be excluded from this study and offered referrals for alcohol treatment.
* Currently seeking or past-12-month history of inpatient or intensive treatment for addictive behaviors
* Psychosis or other severe psychiatric disability
* Pregnancy, nursing or lack of reliable birth control use for women who have not yet reached menopause

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Percent days abstinent via smartphone breathalyzer readings | Baseline to 30 Days
  Within-subject comparison between percent abstinent days based on smartphone breathalyzer readings during the 30-Day Phase 1 Contingency Management induction compared to the 30-day baseline period based on self-report on the timeline followback
Predict percent days abstinent via smartphone breathalyzer readings based on risk factors. | Baseline to 30 Days
  All participants will attempt to reduce alcohol consumption. Only those who are able to will continue to the second phase of the intervention. We will seek to identify which factors are predictive of abstinence.
Perceived value and ease of use of novel contingency management strategies to reduce alcohol consumption. | 30 Days to 60 Days
  Participants will engage in a Contingency Management program aimed at reducing alcohol consumption. A novel CM delivery system will be used intended to gamify the process.
Drinking reduction through Contingency Management will predict non-drinking outcomes | Baseline to 90 days
  Participants who are able to successfully reduce their alcohol consumption may see other health benefits including reduced HIV viral load.

SECONDARY OUTCOMES:
Percent days abstinent via wrist biosensor readings | Baseline to 60 Days
  Among responders during the Phase 1 Contingency Management induction period, comparison among Phase 2 study conditions regarding percent abstinent days based on wrist biosensor readings. Percent days abstinent at baseline based on self-report and based on smartphone breathalyzer readings during Phase 1 will be included in this model.

OTHER OUTCOMES:
Percent days abstinent via self-report | Baseline to 180 Days
  Among responders during the Phase 1 Contingency Management induction period, comparison among Phase 2 study conditions regarding percent abstinent days during the post-intervention, follow-up period based on self-report assessed with the timeline followback from days 61-180. Percent days abstinent at baseline based on self-report and based on smartphone breathalyzer readings during Phase 1 and based on wrist biosensor readings during Phase 2 will be included in this model.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Leeman, Ph.D, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Miami, Coral Gables, Florida
  - University of Florida, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No